CLINICAL TRIAL: NCT04587336
Title: Tailored Approaches to Reduce Distress and Improve Self-Management for Veterans With Diabetes (TARDIS) - Survey & Qualitative Interview
Brief Title: Tailored Approaches to Reduce Distress and Improve Self-Management for Veterans With Diabetes
Acronym: TARDIS
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NRI 18-234
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Diabetes Distress; Self-Management; Veteran
Keywords: Diabetes; Cardiovascular Disease; Self-management; Diabetes Distress; Veteran
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Aim 0 - Cognitive Interview: Examine the understanding and interpretation of diabetes distress and the Diabetes Distress Scale in Veterans with T2D.
  Interventions: Behavioral: Cognitive Interview
- Aim 1 - Baseline Survey: Examine the association of psychosocial factors (depression, PTSD), environmental factors (finances, support), self-management behaviors, and HbA1c with DD.
  Interventions: Behavioral: Baseline Survey; Behavioral: Qualitative Interviews

INTERVENTIONS:
Behavioral: Cognitive Interview — Examine the understanding and interpretation of diabetes distress and the Diabetes Distress Scale in Veterans with T2D.
  Groups: Aim 0 - Cognitive Interview
Behavioral: Baseline Survey — Examine the association of psychosocial factors (depression, PTSD), environmental factors (finances, support), self-management behaviors, and HbA1c with DD.
  Groups: Aim 1 - Baseline Survey
Behavioral: Qualitative Interviews — Describe self-management challenges and preferred learning strategies to inform intervention components and delivery approach for Veterans with T2D.
  Groups: Aim 1 - Baseline Survey

SUMMARY:
Veterans with diabetes may become overwhelmed with the self-management behaviors needed to maintain optimal health. Veterans may experience diabetes distress (DD), a concept distinct from depression, due the amount and frequency of these behaviors. DD negatively influences the Veteran's engagement in self-management and subsequent HbA1c levels. Previous interventions do not tailor T2D self-management information to a Veteran's DD, which may be one reason interventions are ineffective at reducing DD. This proposal examines the impact of correlating factors (e.g., sociodemographic, psychosocial, and environmental) on DD using surveys and semi-structured interviews. This proposal will prepare Allison Lewinski, PhD, MPH, RN for a career as a scientist at VHA focused on developing methods to improve health outcomes among Veterans.

DETAILED DESCRIPTION:
Background: Diabetes self-management is critical to sustaining optimal health following diagnosis. Diabetes distress (DD) is a crucial factor that influences a Veteran's engagement in diabetes self-management. DD is distinct from depression, and includes four domains (i.e., regimen, emotional, interpersonal, healthcare provider). The presence of DD negatively impacts engagement in self-management and HbA1c. Despite interventions aimed at decreasing DD, these interventions have shown minimal lasting effects. One reason may be because interventions do not tailor information to an individual's DD.

Significance & Impact: This proposal will be the first to examine the impact of correlating factors on DD, and then design and test a self-management intervention tailored upon a Veteran's DD type. This proposal addresses the VHA Strategic Plan Priority areas of utilizing resources more efficiently and improving the timeliness of services, and the HSR&D Research Priorities of Population Health/Whole Health and Primary Care Practice. This proposal's findings can improve both care delivery and health outcomes of Veterans, as the investigator will help facilitate the Veteran's linkage to ubiquitous, existing VHA and community services.

Innovation: This proposal will develop an intervention that targets sub-optimal T2D self-management by providing tailored self-management information in conjunction with connections to supportive services. The investigators will identify how, and to what extent, DD and its factors, influence a Veteran's self-management behaviors.

Specific Aims: Aim 1 will examine the association of psychosocial factors (depression, PTSD), environmental factors (finances, support), self-management behaviors, and HbA1c with DD. These Aim 1 data will inform the identification of modifiable factors and selection of the population for a diabetes self-management intervention for Veterans with T2D. Aim 2 will describe self-management challenges and preferred learning strategies to inform the intervention components and delivery approach for Veterans with T2D. Obtaining in-depth perceptions of DD type, self-management strategies and challenges, and learning preferences is essential to tailoring intervention components.

Methodology: This proposal uses an explanatory, sequential mixed-methods design to describe DD in a sample of Veterans who receive care at Durham. In Aim 1 the investigators will survey Veterans (n = 200), and balance enrollment by HbA1C (< 9 or 9) and medication use (insulin, no insulin). In Aim 2 the investigators will conduct semi-structured interviews with a sub-sample (n = ~36) of Veterans surveyed in Aim 1. The investigators will balance enrollment by HbA1C, medication use, and DD level as operationalized by the Diabetes Distress Scale (low, moderate, high).

Implementation & Next Steps: The next steps include dissemination of findings about DD, and its correlates, and the development of an IIR. This IIR will be a Phase III efficacy trial and will be sufficiently powered to test the effects of providing self-management information and connections to supportive services tailored to a Veteran's DD to improve HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes (ICD-10 codes: E11.9, E11.8)
* Documentation of HbA1c drawn within the past 180 days
* Able to speak and read English
* Be able to provide informed consent to participate in the study

Exclusion Criteria:

* New diagnosis of T2D within the last 60 days
* Hospitalization for mental illness within the past 30 days
* Receiving active chemotherapy and/or radiation treatment
* Diagnosis for Metastatic Cancer
* Recent hospitalization within the past 60 days that would influence their diabetes medication regimen (e.g., myocardial infarction, cerebrovascular accident, coronary artery bypass grafting, etc.)
* Currently receiving Kidney Dialysis
* Limited hearing or speech difficulties that influence the Veteran's ability to complete the survey
* Dementia, delirium, or other cognition issues that influence the Veteran's ability to provide consent and complete the survey

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with diagnosis of type 2 diabetes for longer than 60 days with documented HbA1c drawn within 180 days prior to enrollment and able to speak and read English
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lewinski, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewinski AA, Shapiro A, Gierisch JM, Goldstein KM, Blalock DV, Luedke MW, Gordon AM, Bosworth HB, Drake C, Lewis JD, Sinha SR, Husain AM, Tran TT, Van Noord MG, Williams JW Jr. Barriers and facilitators to implementation of epilepsy self-management programs: a systematic review using qualitative evidence synthesis methods. Syst Rev. 2020 Apr 25;9(1):92. doi: 10.1186/s13643-020-01322-9. PMID 32334641
- [Background] Yang Q, Hatch D, Crowley MJ, Lewinski AA, Vaughn J, Steinberg D, Vorderstrasse A, Jiang M, Shaw RJ. Digital Phenotyping Self-Monitoring Behaviors for Individuals With Type 2 Diabetes Mellitus: Observational Study Using Latent Class Growth Analysis. JMIR Mhealth Uhealth. 2020 Jun 11;8(6):e17730. doi: 10.2196/17730. PMID 32525492
- [Background] Lewinski AA, Rushton S, Van Voorhees E, Boggan JC, Whited JD, Shoup JP, Tabriz AA, Adam S, Fulton J, Gordon AM, Ear B, Williams JW Jr, Goldstein KM, Van Noord MG, Gierisch JM. Implementing remote triage in large health systems: A qualitative evidence synthesis. Res Nurs Health. 2021 Feb;44(1):138-154. doi: 10.1002/nur.22093. Epub 2020 Dec 15. PMID 33319411
- [Background] Lewinski AA, Crowley MJ, Miller C, Bosworth HB, Jackson GL, Steinhauser K, White-Clark C, McCant F, Zullig LL. Applied Rapid Qualitative Analysis to Develop a Contextually Appropriate Intervention and Increase the Likelihood of Uptake. Med Care. 2021 Jun 1;59(Suppl 3):S242-S251. doi: 10.1097/MLR.0000000000001553. PMID 33976073
- [Background] Drake C, Batchelder H, Lian T, Cannady M, Weinberger M, Eisenson H, Esmaili E, Lewinski A, Zullig LL, Haley A, Edelman D, Shea CM. Implementation of social needs screening in primary care: a qualitative study using the health equity implementation framework. BMC Health Serv Res. 2021 Sep 17;21(1):975. doi: 10.1186/s12913-021-06991-3. PMID 34530826
- [Background] Lewinski AA, Bosworth HB, Goldstein KM, Gierisch JM, Jazowski S, McCant F, White-Clark C, Smith VA, Zullig LL. Improving cardiovascular outcomes by using team-supported, EHR-leveraged, active management: Disseminating a successful quality improvement project. Contemp Clin Trials Commun. 2021 Feb 6;21:100705. doi: 10.1016/j.conctc.2021.100705. eCollection 2021 Mar. PMID 33644491
- [Background] Lewinski AA, Vaughn J, Diane A, Barnes A, Crowley MJ, Steinberg D, Stevenson J, Yang Q, Vorderstrasse AA, Hatch D, Jiang M, Shaw RJ. Perceptions of Using Multiple Mobile Health Devices to Support Self-Management Among Adults With Type 2 Diabetes: A Qualitative Descriptive Study. J Nurs Scholarsh. 2021 Sep;53(5):643-652. doi: 10.1111/jnu.12667. Epub 2021 Apr 29. PMID 33928755
- [Background] Perez-Aldana CA, Lewinski AA, Johnson CM, Vorderstrasse AA, Myneni S. Exchanges in a Virtual Environment for Diabetes Self-Management Education and Support: Social Network Analysis. JMIR Diabetes. 2021 Jan 25;6(1):e21611. doi: 10.2196/21611. PMID 33492236
- [Background] Rushton S, Lewinski AA, Hwang S, Zullig LL, Ball Ricks KA, Ramos K, Gordon A, Ear B, Ballengee LA, Brahmajothi MV, Moore T, Blalock DV, Williams JW Jr, Cantrell SE, Gierisch JM, Goldstein KM. Barriers and facilitators to the implementation and adoption of improvement coaching: A qualitative evidence synthesis. J Clin Nurs. 2023 Jan;32(1-2):3-30. doi: 10.1111/jocn.16247. Epub 2022 Apr 10. PMID 35403322
- [Background] Ballengee LA, Rushton S, Lewinski AA, Hwang S, Zullig LL, Ricks KAB, Ramos K, Brahmajothi MV, Moore TS, Blalock DV, Cantrell S, Kosinski AS, Gordon A, Ear B, Williams JW Jr, Gierisch JM, Goldstein KM. Effectiveness of Quality Improvement Coaching on Process Outcomes in Health Care Settings: A Systematic Review. J Gen Intern Med. 2022 Mar;37(4):885-899. doi: 10.1007/s11606-021-07217-2. Epub 2022 Jan 3. PMID 34981354
- [Background] Byrd JT, Daniels CL, Flores DD, Kayle M, Lewinski AA, Smith JB, Xu H, Tanabe PJ. Establishing a research racial justice task force to improve diversity, equity, and inclusion in nursing research. Nurs Outlook. 2022 Sep-Oct;70(5):758-761. doi: 10.1016/j.outlook.2022.06.004. Epub 2022 Aug 10. No abstract available. PMID 35961805
- [Background] Lewinski AA, Jazowski SA, Goldstein KM, Whitney C, Bosworth HB, Zullig LL. Intensifying approaches to address clinical inertia among cardiovascular disease risk factors: A narrative review. Patient Educ Couns. 2022 Dec;105(12):3381-3388. doi: 10.1016/j.pec.2022.08.005. Epub 2022 Aug 18. PMID 36002348
- [Background] Lewinski AA, Walsh C, Rushton S, Soliman D, Carlson SM, Luedke MW, Halpern DJ, Crowley MJ, Shaw RJ, Sharpe JA, Alexopoulos AS, Tabriz AA, Dietch JR, Uthappa DM, Hwang S, Ball Ricks KA, Cantrell S, Kosinski AS, Ear B, Gordon AM, Gierisch JM, Williams JW Jr, Goldstein KM. Telehealth for the Longitudinal Management of Chronic Conditions: Systematic Review. J Med Internet Res. 2022 Aug 26;24(8):e37100. doi: 10.2196/37100. PMID 36018711
- [Background] Zullig LL, Lewinski AA, Woolson SL, White-Clark C, Miller C, Bosworth HB, Burleson SC, Garrett MP, Darling KL, Crowley MJ. Research-practice partnerships: Adapting a care coordination intervention for rural Veterans over 3 years at multiple sites. J Rural Health. 2023 Jun;39(3):575-581. doi: 10.1111/jrh.12740. Epub 2023 Jan 20. PMID 36661336
- [Background] German J, Kobe EA, Lewinski AA, Jeffreys AS, Coffman C, Edelman D, Batch BC, Crowley MJ. Factors Associated With Diabetes Distress Among Patients With Poorly Controlled Type 2 Diabetes. J Endocr Soc. 2023 Feb 28;7(5):bvad031. doi: 10.1210/jendso/bvad031. eCollection 2023 Mar 6. PMID 36926446
- [Result] Lewinski AA, Shapiro A, Bosworth HB, Crowley MJ, McCant F, Howard T, Jeffreys AS, McConnell E, Tanabe P, Barcinas S, Coffman CJ, King HA. Veterans' Interpretation of Diabetes Distress in Diabetes Self-Management: Findings From Cognitive Interviews. Sci Diabetes Self Manag Care. 2021 Oct;47(5):391-403. doi: 10.1177/26350106211043487. Epub 2021 Sep 24. PMID 34559032
- [Result] Walsh C, Sullivan C, Bosworth HB, Wilson S, Gierisch JM, Goodwin KB, Mccant F, Hoenig H, Heyworth L, Zulman DM, Turvey C, Moy E, Lewinski AA. Incorporating TechQuity in Virtual Care Within the Veterans Health Administration: Identifying Future Research and Operations Priorities. J Gen Intern Med. 2023 Jul;38(9):2130-2138. doi: 10.1007/s11606-023-08029-2. Epub 2023 Jan 17. PMID 36650326
- [Result] Alexopoulos AS, Soliman D, Lewinski AA, Strawbridge E, Steinhauser K, Edelman D, Crowley MJ. Simplifying therapy to assure glycemic control and engagement (STAGE) in poorly-controlled diabetes: A pilot study. J Diabetes Complications. 2023 Jan;37(1):108364. doi: 10.1016/j.jdiacomp.2022.108364. Epub 2022 Dec 5. PMID 36525906
- [Result] Lian T, Reid H, Rader A, Dewitt-Feldman S, Hezarkhani E, Gu E, Scott M, Kutzer K, Sandhu S, Crowder C, Ito K, Eisenson H, Bettger JP, Shaw RJ, Lewinski AA, Ming DY, Bosworth HB, Zullig LL, Batch BC, Drake C. A Tailored SMS Text Message-Based Intervention to Facilitate Patient Access to Referred Community-Based Social Needs Resources: Protocol for a Pilot Feasibility and Acceptability Study. JMIR Res Protoc. 2022 Oct 11;11(10):e37316. doi: 10.2196/37316. PMID 36222790
- [Result] German J, Yang Q, Hatch D, Lewinski A, Bosworth HB, Kaufman BG, Chatterjee R, Pennington G, Matters D, Lee D, Urlichich D, Kokosa S, Canupp H, Gregory P, Roberson CL, Smith B, Huber S, Doukellis K, Deal T, Burns R, Crowley MJ, Shaw RJ. EXpanding Technology-Enabled, Nurse-Delivered Chronic Disease Care (EXTEND): Protocol and Baseline Data for a Randomized Trial. Contemp Clin Trials. 2024 Nov;146:107673. doi: 10.1016/j.cct.2024.107673. Epub 2024 Aug 30. PMID 39216685
- [Derived] Lewinski AA, Shapiro A, Crowley MJ, Whitfield C, Jones JR, Jeffreys AS, Coffman CJ, Howard T, McConnell E, Tanabe P, Barcinas S, Bosworth HB. Diabetes distress in Veterans with type 2 diabetes mellitus: Qualitative descriptive study. J Health Psychol. 2024 Dec;29(14):1593-1607. doi: 10.1177/13591053241233387. Epub 2024 Feb 21. PMID 38384142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To identify potential participants, we completed computer-based screening using the inclusion/exclusion criteria with medical record data. An informational letter was sent to potential participants and provided contact information if they wanted to opt out. Veterans who did not opt out were screened for eligibility using a telephone-based screening questionnaire. Participants were recruited from August 2020 - July 2021 for the surveys and cognitive interviews.
Pre-assignment Details: Participants who are listed under started for the time periods below were only enrolled/consented to participate and were not assigned an intervention at that time point. All participants have the option to voluntarily withdraw at any time during the study period. Participants who completed study procedures (baseline cognitive interview or baseline survey) were noted as completed within the participant flow.
Groups:
- Aim 0 - Cognitive Interview: Cognitive Interviews: Examine the understanding and interpretation of diabetes distress and the Diabetes Distress Scale in Veterans with T2D.
  Cognitive Interview: Cognitive Interviews: Examine the understanding and interpretation of diabetes distress and the Diabetes Distress Scale in Veterans with T2D.
- Aim 1 - Baseline Survey: Conduct Baseline Survey: Examine the association of psychosocial factors (depression, PTSD), environmental factors (finances, support), self-management behaviors, and HbA1c with DD.
  Baseline Survey: Conduct Baseline Survey: Examine the association of psychosocial factors (depression, PTSD), environmental factors (finances, support), self-management behaviors, and HbA1c with DD.
  Qualitative Interviews: Qualitative Interviews: Describe self-management challenges and preferred learning strategies to inform intervention components and delivery approach for Veterans with T2D.
Period: Overall Study
Arm/Group | Aim 0 - Cognitive Interview | Aim 1 - Baseline Survey
Started | 15 | 210
Completed | 14 | 210
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aim 0 - Cognitive Interview | Aim 1 - Baseline Survey | Total
Number analyzed (Participants) | 15 | 210 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.867 (8.551) | 63.386 (10.235) | 63.218 (10.134)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 32 | 36
  Male | 11 | 178 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 8
  Not Hispanic or Latino | 15 | 202 | 217
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 128 | 136
  White | 6 | 65 | 71
  More than one race | 1 | 7 | 8
  Unknown or Not Reported | 0 | 5 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 210 | 225

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: Differences in Diabetes Distress Scale Score by HbA1c Level (HbA1c < 9 and HbA1c ≥ 9)
Description: Scale used: 17 item Diabetes Distress Scale. Minimum value 1, Maximum value 6 Scoring is: < 2.0 is little or no distress; 2.0-2.9 is moderate distress; and ≥ 3.0 is high distress.
  Higher scores indicate higher diabetes distress or worse outcome.
Time Frame: Baseline
Population: Veterans are classified into well-controlled (defined by HbA1c value < 9 during the past 180 days) and poorly-controlled (HbA1c value ≥ 9 during the past 180 days).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- HbA1c < 9: HbA1c < 9 represents well-controlled type 2 diabetes (defined by HbA1c value < 9 during the past 180 days).
- HbA1c ≥ 9: HbA1c ≥ 9 represents poorly-controlled type 2 diabetes (defined by HbA1c value ≥ 9 during the past 180 days).
Arm/Group | HbA1c < 9 | HbA1c ≥ 9
Number analyzed (Participants) | 109 | 101
score on a scale | 1.907 (0.882) | 2.054 (0.943)

2. Primary Outcome: Aim 1: Differences in Diabetes Distress Scale Score by Medication Regimen (no Insulin, Insulin).
Description: Scale used: 17 item Diabetes Distress Scale. Minimum value 1, Maximum value 6 Scoring is: < 2.0 is little or no distress; 2.0-2.9 is moderate distress; and ≥ 3.0 is high distress Higher scores indicate higher diabetes distress or worse outcome.
Time Frame: Baseline
Population: Veterans are classified into no insulin (defined by taking only oral T2D medications and/or non-insulin injectable medications during the past 180 days) and insulin (defined by taking any insulin during the past 180 days; these Veterans may/may not also take oral T2D medication(s)).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Insulin: Defined by taking any insulin during the past 180 days; these Veterans may/may not also take oral T2D medication(s)
- No Insulin: Defined by taking only oral T2D medications and/or non-insulin injectable medications during the past 180 days
Arm/Group | Insulin | No Insulin
Number analyzed (Participants) | 117 | 93
score on a scale | 2.102 (1.013) | 1.824 (0.749)

ADVERSE EVENTS:
Time Frame: Baseline
Arm/Group | Aim 0 - Cognitive Interview | Aim 1 - Baseline Survey
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/210
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/210
Other Adverse Events (participants affected / at risk) | 0/15 | 0/210

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT04587336/Prot_SAP_000.pdf